CLINICAL TRIAL: NCT02152683
Title: Linear Focused Shockwave Treatment for Erectile Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Initia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LISW-NY
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2015-09

CONDITIONS: Vasculogenic Erectile Dysfunction

ARMS (2):
- long protocol (Experimental): Renova
  Interventions: Device: Renova
- short protocol (Experimental): Renova
  Interventions: Device: Renova

INTERVENTIONS:
Device: Renova — Low- Intensity Shockwave

SUMMARY:
The study is aimed at comparing the performance of protocols employing one and two sessions per week, respectively. The study hypothesis claims that there is no significant difference between the performances of the compared protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health
2. Vasculogenic ED- Erectile Dysfunction, according to physician judgment, for at least 6 months and for no longer than 5 years.
3. International Index of Erectile Function 6 (IIEF-EF) between 17 and 25
4. Satisfactory response to the use of PDE5 (Phosphodiesterase type 5) inhibitors
5. Stable sexual relationship for at least 3 months prior to treatment
6. Minimum of two sexual attempts per month

Exclusion Criteria:

1. Hormonal, neurological or psychological pathology
2. Past radical prostatectomy or extensive pelvic surgery
3. Recovering from cancer during last year
4. Any unstable medical, psychiatric, spinal cord injury and penile anatomical abnormalities
5. Clinically significant chronic hematological disease
6. Anti-androgens, oral or injectable androgens
7. Past radiotherapy treatment of the pelvic region
8. International normalized ratio (INR) > 3 for patients using blood thinners (such as Coumadin)

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
IIEF-EF- International Index of Erectile Function questionnaire score | 1 month post treatment
  the IIEF-EF questionnaire score will be evaluated at baseline, 1,3, and 6 months after end of treatment
IIEF-EF questionnaire score | 3 months post treatment
IIEF-EF questionnaire score | 6 months post treatment
  the IIEF-EF questionnaire score will be evaluated at baseline, 1,3, and 6 months after end of treatment

SECONDARY OUTCOMES:
SEP- Sexual Encounter Profile: Questions 2 and 3 | 1, 3 and 6 months post treatment
GAQ- Global Assessment Questions | 1, 3 and 6 months post treatment
EHS- Erection Hardness Score | 1, 3 and 6 months post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Eastchester Center for Cancer Care, New York, New York, United States

REFERENCES:
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Goyal NK, Garg M, Goel A. Re: Does low intensity extracorporeal shock wave therapy have a physiological effect on erectile function? Short-term results of a randomized, double-blind, sham controlled study: Y. Vardi, B. Appel, A. Kilchevsky and I. Gruenwald. J Urol 2012; 187: 1769-1775. J Urol. 2012 Nov;188(5):2018-9. doi: 10.1016/j.juro.2012.07.052. Epub 2012 Sep 20. No abstract available. PMID 22999553
- [Background] Rosen RC, Cappelleri JC, Gendrano N 3rd. The International Index of Erectile Function (IIEF): a state-of-the-science review. Int J Impot Res. 2002 Aug;14(4):226-44. doi: 10.1038/sj.ijir.3900857. PMID 12152111
- [Background] Rosen RC, Allen KR, Ni X, Araujo AB. Minimal clinically important differences in the erectile function domain of the International Index of Erectile Function scale. Eur Urol. 2011 Nov;60(5):1010-6. doi: 10.1016/j.eururo.2011.07.053. Epub 2011 Jul 30. PMID 21855209